CLINICAL TRIAL: NCT05163301
Title: Alcohol Research Consortium in HIV: Relapse Prevention Arm
Brief Title: Alcohol Research in HIV: Relapse Prevention
Acronym: ARCH-RPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00288483
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: HIV; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: one group will receive computer delivered relapse prevention intervention (RPI); one group will receive person delivered relapse prevention intervention; one group will receive usual care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computer delivered RPI (Experimental): 2 session computer delivered counseling to prevent relapse to hazardous drinking
  Interventions: Behavioral: Relapse Prevention Intervention
- Person delivered RPI (Experimental): 2 session counselor delivered counseling to prevent relapse to hazardous drinking
  Interventions: Behavioral: Relapse Prevention Intervention
- Treatment as Usual (No Intervention): Counseling for alcohol use available in clinic as treatment as usual

INTERVENTIONS:
Behavioral: Relapse Prevention Intervention — 2 session intervention to address relapse prevention among people with HIV who have an alcohol use disorder
  Arms: Computer delivered RPI; Person delivered RPI

SUMMARY:
3-arm type 1 pilot implementation-efficacy trial for people with alcohol use disorders to examine the preliminary effectiveness and feasibility of an adapted 2-session, computerized and person delivered relapse prevention intervention.

DETAILED DESCRIPTION:
This study will develop a brief counseling intervention for people with HIV who have resumed alcohol use or resumed hazardous alcohol use after a minimum of 3 years of alcohol abstinence or 'lower risk' alcohol use. The investigators will develop a 2session person delivered and a 2-session computer delivered intervention which the investigators will then compare with the usual treatment for alcohol counseling offered at the HIV clinic. The investigators will also study the acceptability and feasibility of implementing both types of counseling in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HIV
* Aged 18 years or older
* Must be enrolled in clinical care at Johns Hopkins HIV Clinic.

In addition, meet the following alcohol use criteria:

1. lifetime alcohol use disorder
2. patient reported outcomes (PRO) assessment collected by the Center for AIDS Research (CFAR) Network of Clinical Systems as part of usual clinical care that show in the last 3 years: periods of no or lower risk drinking (e.g. women/men who are drinking <11/22 drinks per week) and periods of lapse to higher levels of drinking (=>11/22 drinks per week for women/men)
3. current PRO showing alcohol abstinence or alcohol use at <11/22 drinks per week for women/men.

Exclusion Criteria:

* Acutely suicidal, homicidal, psychotic or otherwise unable to provide informed consent
* Non-English speaking because interventions are currently available in English only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in time to relapse | 6 and 12 months
  Time to return to any alcohol use or any at risk alcohol use after intervention.

SECONDARY OUTCOMES:
Alcohol use pattern as assessed by change in number of drinking days | Baseline, 6 and 12 months
  Number of drinking days.
Alcohol use pattern as assessed by change in number of heavy drinking days | Baseline, 6 and 12 months
  Number of heavy drinking days.
Alcohol use pattern as assessed by change in number of drinks per drinking day | Baseline, 6 and 12 months
  Number of drinks per drinking day.
Alcohol use pattern as assessed by change in number of days abstinent | Baseline, 6 and 12 months
  Number of days abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Hutton, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NIAAA has begun a new data-sharing initiative to create a data repository of future NIAAA-funded studies that include human subjects. This repository is called the NIAAA Data Archive (NIAAA DA). NIAAA-funded investigators conducting human subjects research are expected to submit de-identified, individual-level data to this data archive.
  The NIAAA DA accepts only electronic, de-identified data from human subjects studies. Data submitted to the NIAAA DA must be de-identified by the investigator prior to submission.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared with the general research community 2 years after the grant end date on the initial Notice of Award. This 2-year embargo period will provide study investigators with protected time to publish from the study data. After the embargo, the data will be made available for sharing with the general research community via the NIAAA DA website. However, if a manuscript using study data is accepted for publication prior to the 2-year embargo, the study data specifically used in that manuscript will be shared with the general research community at the time of publication.
Access Criteria: Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NIAAA DA data by submitting a data access request in accordance with applicable NIAAA DA policies. Data requests will be reviewed and granted by a NIAAA Data Access Committee.
URL: https://grants.nih.gov/grants/guide/notice-files/NOT-AA-19-020.html